CLINICAL TRIAL: NCT06943404
Title: Prevention/Reduction of ASRs and PTSD to Sustain Civilian Performance With a Sublingual Formulation of Dexmedetomidine (BXCL501)
Brief Title: BXCL501 After Stress to Increase Recovery Success
Acronym: RISE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Mclean Hospital (Other); Washington University School of Medicine (Other); University of Florida (Other); Rhode Island Hospital (Other); Vanderbilt University School of Medicine (Other); Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 25-0345
Record Dates: First submitted 2025-04-15; First posted 2025-04-24 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Acute Stress Reaction; Acute Stress Disorder; Post-traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Traumatic, Acute; Stress Disorders, Post-Traumatic | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BXCL501 (dexmedetomidine HCl) (Experimental): Participants will be instructed to take an initial dose of BXCL501 (equivalent to 1 film, 120mcg) in the ED as part of enrollment procedures. If the time between the first dose and the planned bedtime of the participant is greater than 6 hours, participants will be instructed to take the second dose at bedtime on the day of enrollment. If the time between the first dose and the planned bedtime of the participant is less than 6 hours participants will be instructed to take the second dose before bedtime on the day following enrollment. Following the initial dosing on the day of enrollment, all participants will be instructed to take a dose of study medication before bedtime until they have completed 14 days of treatment.
  Interventions: Drug: BXCL501 (dexmedetomidine HCl)
- Placebo (Placebo Comparator): Participants will be instructed to take an initial dose of placebo (equivalent to 1 film, 120mcg) in the ED as part of enrollment procedures. If the time between the first dose and the planned bedtime of the participant is greater than 6 hours, participants will be instructed to take the second dose at bedtime on the day of enrollment. If the time between the first dose and the planned bedtime of the participant is less than 6 hours participants will be instructed to take the second dose before bedtime on the day following enrollment. Following the initial dosing on the day of enrollment, all participants will be instructed to take a dose of study medication before bedtime until they have completed 14 days of treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BXCL501 (dexmedetomidine HCl) — BXCL501 (dexmedetomidine HCl) taken sublingually (under the tongue) in the ED and at bedtime over 2 weeks.
  Other Names: BXCL501
  Arms: BXCL501 (dexmedetomidine HCl)
Drug: Placebo — Placebo taken sublingually (under the tongue) in the ED and at bedtime over 2 weeks.
  Arms: Placebo

SUMMARY:
This study will examine the safety and efficacy of BXCL501 to reduce ASR symptoms and behavioral changes among patients presenting to the Emergency Department (ED) after Motor Vehicle Collision (MVC). Specifically, the investigators will perform the BXCL501 (BASIS) Trial, a double-blind placebo-controlled Randomized Controlled Trial (RCT) to determine if BXCL501 (dexmedetomidine hydrochloride sublingual film) initiated in the ED in the hours after MVC to high risk individuals, treats/reduces ASR/ASD symptoms (primary outcome), improves neurocognitive function, and prevents/reduces posttraumatic stress (PTS) symptoms (secondary outcomes) long term. 100 participants will be randomized, receive study drug in ED and be discharged with a 2-week drug supply. Prior to initial dose of study drug administration, and during the hours, days, and weeks after participants will receive serial longitudinal assessments of psychological and somatic symptoms, neurocognitive function, and adverse events.

DETAILED DESCRIPTION:
U.S. military personnel are exposed to life-threatening traumatic events (e.g., intense firefights with multiple casualties) that result in acute stress reaction (ASR) symptoms (ICD-10) and posttraumatic stress (PTS). Similarly, acute and persistent stress symptoms, and related adverse posttraumatic neuropsychiatric sequelae, are also very common and cause a tremendous burden of suffering in civilian populations following exposure to life-threatening traumatic events (e.g., motor vehicle collision, violent or accidental death of a loved one, and assault). BXCL501 (dexmedetomidine HCl sublingual film) has been evaluated in multiple clinical trials across a range of medical conditions (dementia, schizophrenia, bipolar disorder, opioid use disorder), with an excellent safety profile, and evidence of efficacy with respect to decreasing agitation. This is promising for the treatment of ASRs, as agitation is a primary feature of ASRs in many individuals. Additionally, adrenergic hyperactivity is also a key characteristic of ASRs and contributes to the development of Posttraumatic Stress Disorder (PTSD). BXCL501 is known to decrease the activity of central noradrenergic neurons, suggesting a mechanistic pathway by which BXCL501 may improve outcomes for individuals at risk of ASR/ASD/PTSD. BXCL501 therefore holds significant promise as a treatment aimed at reducing ASR symptoms and related behavioral changes, enhancing resilience and improving warfighter performance, and reducing the frequency and severity of persistent/chronic PTS symptoms. This study will evaluate the safety and efficacy of BXCL501 in a population of trauma survivors at high risk for developing ASR, ASD, and PTSD symptoms, and may ultimately provide military personnel, veterans, and civilians with an important new treatment option to improve recovery, job performance, and quality of life when administered in the early aftermath of exposure to a traumatic stressor.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years and ≤ 65 years of age
* Admitted to ED within 24 hours of MVC
* Anticipated to be discharged home from the ED
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Consent to receive unencrypted communications
* Has a smartphone with continuous service for more than 1 year
* Has a personal email address they regularly access
* Able to speak and read English
* Females of childbearing potential (not surgically sterilized (tubal ligation/hysterectomy) or not post-menopausal (no menstrual period for > 12 months)) must be willing to use a medically acceptable and effective birth control method for 3 months before the study and while participating in the study. Medically acceptable methods of contraception that may be used by the participant include abstinence, birth control pills or patches, birth control implants, diaphragm, intrauterine device (IUD), or condoms.

Exclusion Criteria:

* Substantial comorbid injury (e.g., long bone fracture)
* People of childbearing potential who are pregnant, breastfeeding, planning to become pregnant, or not using a highly effective form of contraception (e.g., implants, intrauterine devices (IUDs), tubal ligation, hormonal birth control pills, patches, vaginal rings, or injections) during their participation
* Prisoner status
* Chronic daily opioid use prior to MVC (> 20 mg oral daily morphine equivalents)
* Bipolar disorder, psychotic disorder, active psychosis, suicidal ideation, or homicidal ideation
* Hospital admission
* Clinically significant history of cardiac disease including (a) history of syncope or other syncopal attacks; (b) current evidence of orthostatic hypotension (defined as a decrease in systolic BP of 20 mm Hg or decrease in diastolic BP of 10mm Hg within 3 minutes); (c) resting heart rate of <55 beats per minute; (d) systolic blood pressure <110mmHg or diastolic BP <70mmHg; or (e) participants with a QTC interval >440msec (males) or >460msec (females) not in sinus rhythm; or 1st, 2nd or 3rd degree hearth block
* Hypomagnesia (<1.7 mg/dL)
* Substantial hepatic impairment (AST or ALT > 3 times the upper limit of normal).
* Currently taking the following medications: a) medications for alcoholism (e.g. naltrexone, disulfiram, topiramate, acamprosate); b) psychotropic medications that promote sedation including sedative/hypnotics, barbiturates, antihistamines, sedative antidepressants (e.g. doxepin, mirtazapine, trazodone), and triptans (e.g., sumatriptan); c) alpha-2-adrenergic agonists (clonidine, guanfacine, lofexidine); d) adrenergic agents prescribed for other reasons (prazosin); e) or medications known to cause QT prolongation.(Permitted Concomitant Medications: The concomitant medications allowed in the study include non-sedative antidepressants used to treat PTSD)
* Hypersensitivity or history of allergic reaction to dexmedetomidine
* Lacking capacity to provide informed consent (receipt of sedative, hypnotic agent making the patient non-decisional for consent)
* Any other history or condition that would, in the site investigator's judgement, indicate that the patient would very likely be non-compliant with the study or unsuitable for the study (e.g., might interfere with the study, confound interpretation, or endanger patient)
* Participation in any other clinical trial of a pharmacological agent within 30 days prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-02-11 (Estimated); Primary Completion 2026-09-29 (Estimated); Study Completion 2026-09-29 (Estimated)

PRIMARY OUTCOMES:
Change in ASD Score | Week 1, 3 after MVC
  Individuals are asked to complete the 14-item Acute Stress Disorder Scale (ASDS) self-report inventory where each item is rated on a 5-point scale (0= Not at all; 1= Mildly; 2= Medium; 3= Quite a bit; 4= Very Much) that indexes acute stress disorder (ASD). Range of possible total scores is 0-56, with higher total scores indicating greater acute stress symptoms.

SECONDARY OUTCOMES:
Median reaction time of correct responses (general cognitive function) | Min 30, Hour 1, 6, 12, Day 1, 2, 3, Week 1, 2, 3, 5, 6, 8, 11, 12 after MVC
  General cognitive function will be assessed using the Test My Brain Digit Symbol Matching Test. Participants will be asked to match symbols and numbers using a symbol-number key shown on screen. General cognitive function is assessed via measuring median reaction time of correct responses (medianRTc) to 'test' trials. Range for medianRTc (ms) is 0-30000.
Median reaction time of correct responses (procedural reaction time) | Min 30, Hour 1, 6, 12, Day 1, 2, 3, Week 1, 2, 3, 5, 6, 8, 11, 12 after MVC
  Procedural reaction time will be assessed using the Test My Brain Choice Reaction Time Test. Participants see a set of three arrows, where one arrow is a different color from the rest. The participant presses left or right to indicate the direction of the odd colored arrow. Reaction time is assessed via measuring median reaction time of correct responses (medianRTc) to 'test' trials. Range for medianRTc (ms) is 0-5000.
Proportion of targets correctly identified (visuospatial processing and attention) | Min 30, Hour 1, 6, 12, Day 1, 2, 3, Week 1, 2, 3, 5, 6, 8, 11, 12 after MVC
  Visuospatial processing and attention will be assessed using the Test My Brain Multiple Object Tracking Test. In this test of visuospatial processing and attention, participants have to track a set of target circles around the screen (amidst a field of distractors) that move at increasing speed with each trial. Once the circles stop moving, participants select which were targets must identify targets instead of distractors. Visuospatial processing and attention are assessed via the proportion of targets correctly identified. Range for measure is 0-1.
d-prime identification (psychomotor vigilance) | Min 30, Hour 1, 6, 12, Day 1, 2, 3, Week 1, 2, 3, 5, 6, 8, 11, 12 after MVC
  Psychomotor vigilance will be assessed via the Test My Brain Gradual Onset Continuous Performance Test. In this task, participants monitor a stream of city and mountain images that rapidly fade from one to the next with no interstimulus interval. Participants are asked to press/touch for each city image and to withhold for each mountain image. Vigilance is assessed via measuring d-prime for identification of each city image, a signal detection-based measure that takes into account both hits and false alarms to provide an unbiased estimate of performance where higher values reflect better performance. Response inhibition is defined as the suppression of actions that are inappropriate in a given context. Response inhibition is assessed using results from the above, by measuring the number of commission errors (failure to withhold responses) where most positive scores reflect more impulsive responding. Range for measure is -4.2279 to 4.2279.
Change in Pain Symptom Score | Baseline, Week 1, 3, 6, 12 after MVC
  The Regional Pain Scale (RPS) will be used to assess the extent of body pain. 13 items will be scored on a 0-10 pain scale where 0 is no pain and 10 is severe pain. Range of possible total scores is 0-130, with higher total scores indicative of greater pain symptoms
Change in Depressive Symptoms Score | Baseline, Week 1, 3, 6, 12 after MVC
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Depression Short Form 8b; an 8-item scale, and one question from the PROMIS Depression Item Bank will be aggregated/combined to assess depression. Each item is scored on a 5-point scale where 0 is "none of the time" and 5 means "all or almost all of the time". Range of possible total scores is 0-45, with higher total scores indicative of greater depressive symptoms.
Change in Somatic Symptom Score | Baseline, Week 1, 3, 6, 12 after MVC
  The Pennebaker Inventory of Limbic Languidness (PILL) assesses the frequency of common physical symptoms and sensations. The investigators will use a version with adapted response options for greater consistency across measures, greater precision in response levels, and to allow administration via self-report. 20 items will be scored on a 0-10 scale where 0 is "no problem" and 10 means "major problem". Range of possible total scores is 0-200, with higher total scores indicative of greater somatic symptoms.
Change in PTSD Symptoms | Baseline, Week 1, 3, 6, 12 after MVC
  The PTSD Checklist for DSM-5 (PCL-5) assesses PTSD symptoms as defined by the Diagnostic and Statistical Manual of Mental Disorders-5th Edition (DSM-5). 20 items will be scored on a five-point scale ranging from 0 ("not at all") to 4 ("extremely"). Range of possible total scores is 0-80, with higher total scores indicative of greater PTSD symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel McLean, MD, Principal Investigator — University of North Carollina at Chapel Hill; Stacey House, MD, Principal Investigator — Washington University School of Medicine
Locations (3):
- United States (3):
  - University of Florida College of Medicine - Jacksonville, Jacksonville, Florida
  - Washington University in St. Louis, St Louis, Missouri
  - UVA University Hospital, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 12 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with University of North Carolina at Chapel Hill (UNC).
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 12 months following publication and continuing for 36 months.
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.